CLINICAL TRIAL: NCT00719966
Title: Effect of Aromatase Inhibitor Therapy for Breast Cancer on Endothelial Function
Brief Title: Effect of Aromatase Inhibitor Therapy on Blood Vessel Function in Postmenopausal Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MC0834; 06-004006 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Anastrozole; exemestane; Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 (hormone receptor-positive): Patients receive aromatase inhibition therapy for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: anastrozole; Drug: exemestane; Drug: letrozole; Procedure: assessment of therapy complications
- Group 2 (hormone receptor-negative): Patients do not receive adjuvant treatment.
  Interventions: Procedure: assessment of therapy complications

INTERVENTIONS:
Drug: anastrozole — Patients receive aromatase inhibition therapy.
  Groups: Group 1 (hormone receptor-positive)
Drug: exemestane — Patients receive aromatase inhibition therapy.
  Groups: Group 1 (hormone receptor-positive)
Drug: letrozole — Patients receive aromatase inhibition therapy.
  Groups: Group 1 (hormone receptor-positive)
Procedure: assessment of therapy complications — Endothelial function is measured

SUMMARY:
RATIONALE: Aromatase inhibitor therapy is used in treating postmenopausal women who have hormone-dependent breast cancer. It is not yet known what effect aromatase inhibitor therapy has on blood vessel function.

PURPOSE: This clinical trial is studying the effect of aromatase inhibitor therapy on blood vessel function in postmenopausal women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of adjuvant aromatase inhibitor therapy on endothelial function in postmenopausal women with breast cancer.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 treatment groups according to breast cancer hormone-receptor status (positive vs negative).

* Group 1 (hormone receptor-positive): Patients receive aromatase inhibition therapy for up to 6 months in the absence of unacceptable toxicity.
* Group 2 (hormone receptor-negative): Patients do not receive adjuvant treatment.

Endothelial function is measured in both groups at baseline and at follow up by the room temperature peripheral arterial tonometry (RT-PAT) index using the EndoPAT method.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Ductal carcinoma in situ (DCIS) allowed provided the patient will not receive tamoxifen as part of treatment for their cancer
* May not have had a prior mastectomy with requirement for mastectomy of the contralateral breast
* No requirement for axillary lymph node dissection with a history of contralateral mastectomy and/or contralateral axillary lymph node dissection
* Hormone receptor status meeting 1 of the following criteria:

  * Hormone receptor negative and not eligible for aromatase inhibitor therapy (AI)
  * Hormone receptor positive and are not receiving an AI

PATIENT CHARACTERISTICS:

* Postmenopausal
* No known or symptomatic coronary artery disease
* No significant co-morbidities, including any of the following conditions:

  * Active renal or hepatic disease
  * Known uncontrolled and/or untreated peripheral arterial disease
  * Uncontrolled and/or untreated hypertension
  * Uncontrolled and/or untreated diabetes
  * Uncontrolled and/or untreated hyperlipidemia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 7 days since prior hormone replacement therapy or hormone-based contraception
* More than 12 months since prior and no concurrent tamoxifen or aromatase inhibitor therapy for this disease
* More than 12 months since prior and no concurrent chemotherapy for this disease
* No prior bilateral mastectomy

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recently diagnosed breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2008-09-18 (Actual); Primary Completion 2013-06-13 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Endothelial dysfunction as a result of aromatase inhibitor therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nicole P. Sandhu, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States